CLINICAL TRIAL: NCT01253252
Title: Endoprosthesis Treatment Effects on Human Abdominal Aorta Aneurysms(AAA)Metabolic Activity
Brief Title: Endoprosthesis Treatment Effects on Human Abdominal Aorta Aneurysms (AAA) Metabolic Activity
Acronym: AAAendo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-A01424-49
Record Dates: First submitted 2010-02-05; First posted 2010-12-03 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; Prosthesis; Fluorodeoxyglucose F18; Positron-emission Tomography; Spiral computed tomography; Biological markers
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Specific procedure (Experimental): A [18F] Fluorodeoxyglucose PET Scan Imaging will be added to their conventional follow up (CT scan, usual blood sampling, ECG…) i.e. within one month before endovascular surgery (inclusion visit), at one month and 6 month of follow-up.
  Furthermore, blood sampling for biological investigations (biological markers of the inflammation, proteolysis and coagulation potentially related to morphology and evolution of AAA) will be done.
  Interventions: Radiation: [18F] Fluorodeoxyglucose PET Scan Imaging; Radiation: CT scan; Biological: Blood sampling for biological investigations

INTERVENTIONS:
Radiation: [18F] Fluorodeoxyglucose PET Scan Imaging — Positron Emission Tomography (PET) is a nuclear medicine imaging technique which produces a 3-dimensional image of functional processes in the body. The system detects pairs of gamma rays emitted indirectly by a positron-emitting radionuclide, which is introduced into the body on a biologically active molecule. Images of tracer concentration in 3-dimensional space are then reconstructed by computer analysis.
  The biologically active molecule chosen for PET is 18-fluorodeoxyglucose. The concentrations of tracer imaged then give tissue metabolic activity, in terms of regional glucose uptake.
  The dose of 18FDG that is recommended for adults in a standard exploration varies from 200 to 500 MBq according to the weight of the patient and the camera used. No allergic or other incident has been observed after several thousands of examinations.
Radiation: CT scan — Computed tomography (CT) is a medical imaging method employing tomography created by computer processing. Digital geometry processing is used to generate the PET's three-dimensional space image.
Biological: Blood sampling for biological investigations — A venous blood sample of a total of 30 ml for measurement of enzymes associated with the development of aneurysms (= biomarkers).

SUMMARY:
The purpose of this study is to determine whether Positron Emission Tomography imaging can help to predict the evolutivity of AAA treated with endovascular prosthesis.

DETAILED DESCRIPTION:
Background:

Abdominal Aorta Aneurysm(AAA) is a frequently occurring atherothrombotic disease, linked to male gender and aging. Due to the current aging of the population, the incidence of rupture may be increasing. The clinical evaluation of AAA usually includes a morphological assessment(size and localization) for diagnosis, open surgery or endovascular prosthesis (EVAR) may be indicated to prevent the onset of a rupture which is often lethal. Unfortunately, the durability of endovascular repair of AAA remains uncertain and the rupture risk or endoleaks onset requires continuous surveillance and the conventional imaging by CT scan often fails to predict this negative progression.

Our hypothesis is that the therapeutic efficacity of endovascular surgery in the AAA is linked to the restoration of effective compartmentalization between the blood and the outer wall (removal of the thrombosis interface and blood pressure constraint). Thus, success of EVAR must be followed by the disappearance of adventitial inflammation visualized by metabolic activity in FDG-PET (18FDG uptake) and a normalization of biological markers of the injury. Conversely, the inefficacy of endovascular therapy should result in the persistence of an inflammatory metabolic activity in relation to the saccular endoleak and a persistent elevation of plasma biomarkers.

Primary objective:

The general aim of this pilot study is to assess the effect of endoprosthesis treatment on PET scan functional imaging of AAA.

Materials and method:

Seven French Hospitals will recruit 50 patients presenting a large AAA scheduled for EVAR (Endovascular prosthesis) within one month. A 18FDG PET scan will be added to their conventional follow up (CT scan, usual blood sampling, ECG…) i.e. within one month before endovascular surgery (inclusion visit), at one month and 6 month of follow-up.

Furthermore, biological markers of the inflammation, proteolysis and coagulation potentially related to morphology and evolution of AAA will be investigated by the U698 (National Institute for Medical Research) Unit, implementing already existing database from others cohorts of patients with AAA, including biological samples conserved both by the Nancy clinical investigation center and the (U698) National Institute for Medical Research Unit.

Study duration for a patient: 26 months

Perspectives:

This pilot study will help to assess the effect of EVAR in terms of it functional inflammatory response and determine the required sample size for a future project. Since aneurysm expansion rate varies widely among patients and even for one single patient over time, studying metabolic adventitial immuno-inflammatory activity using 18FDG PET imaging will provide new major informations about the efficacity of endovascular therapy in AAA. Plasma assays will help to identify intermediate biological markers of aneurysm evolutivity after endovascular therapy. Those complementary functional and biological criteria are of paramount importance to improve therapeutic management and prognosis of AAA.

ELIGIBILITY:
Inclusion Criteria:

* Large AAA scheduled for endovascular surgery within one month
* Written informed consent

Exclusion Criteria:

* Evolutive neoplasm
* Chronic liver disease
* Connective tissue diseases: rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, Crohn's disease, polymyositis/dermatomyositis, mixed connective tissue disease
* Crohn's disease
* Evolutive tuberculosis
* Contraindication to CT scan
* Pregnancy and breastfeeding
* Women of child bearing potential
* Patient unable to understand the study aims
* Patient unable to comply with scheduled visit
* Participation in other investigational studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Difference of 18FDG PET scan signal (mean and maximal aortic standardized uptake measurements) visualized before and after endoprosthesis implantation for AAA treatment. | 3 Pet scan will be performed: within one month before surgery and after 1 and 6 months of follow-up

SECONDARY OUTCOMES:
Correlation between therapeutic efficacity of endovascular treatment and AAA injury biological markers. | Blood samplings will be performed 5 times: within one month before endoprosthesis implantation and after one month, six months, one year and 2 years of follow-up
Relationship between efficacity of endovascular surgery and morphology of the AAA as assessed by CT scan. | CT scan will be performed within one month before endoprosthesis implantation and at one month, six months, one year and two years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Patrick ROSSIGNOL, MD, phD, Principal Investigator — Nancy's Hospital, Plurithematic Clinical Investigation Centre; Jean-Baptiste MICHEL, MD, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale (INSERM) U698 FRANCE
Locations (7):
- France (7):
  - Le Bocage - Dijon's Hospital, Dijon
  - Cardiologic Hospital, Lille
  - Brabois Hospital, Nancy
  - Institut du Thorax, Nantes's Hospital, Nantes
  - Bichat Claude Bernard Hospital, Paris
  - Georges Pompidou European Hospital, Paris
  - CH.NICOLLE's Hospital, Rouen